CLINICAL TRIAL: NCT00996723
Title: Phase I Study of the Combination of Vandetanib and Dasatinib Administered During and After Radiation Therapy in Children With Diffuse Intrinsic Pontine Glioma
Brief Title: Clinical Trial Evaluating the Combination of Vandetanib and Dasatinib During and After Radiation Therapy (RT) in Children With Newly Diagnosed Diffuse Intrinsic Pontine Glioma (DIPG)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: AstraZeneca (Industry); The Cure Starts Now Foundation (Unknown); Tyler's Treehouse (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SJBG09; NCI-2011-01152 (Registry Identifier: NCI Clinical Trial Registration Program)
Record Dates: First submitted 2009-10-15; First posted 2009-10-16 (Estimated); Last update posted 2015-04-06 (Estimated); Status verified 2015-04

CONDITIONS: Diffuse Intrinsic Pontine Glioma
MeSH Terms: conditions — Diffuse Intrinsic Pontine Glioma | interventions — vandetanib; Dasatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Other)
  Interventions: Drug: vandetanib and dasatinib

INTERVENTIONS:
Drug: vandetanib and dasatinib — Two oral investigational agents (vandetanib [VEGFR2, RET, and EGFR inhibitor] and dasatinib [bcr-abl, PDGFRA and B, src, lck, yes, and c-kit inhibitor] will be administered during and after local RT, which is the only standard therapy for children with DIPG.

SUMMARY:
This is a Phase I clinical trial evaluating the combination of vandetanib and dasatinib during and after radiation therapy (RT) in children with newly diagnosed diffuse intrinsic pontine glioma (DIPG).

DETAILED DESCRIPTION:
This trial will estimate the maximum safe dose of vandetanib and dasatinib which can be administered during the 6 weeks of local RT in children with newly diagnosed DIPG.

ELIGIBILITY:
Inclusion Criteria:

1. Age must be ≥ 18 months and < 21 years
2. Diagnosis of DIPG or high-grade glioma originating from the brainstem.
3. Lansky (for research participants ≤ 16 years) or Karnofsky (for research participants > 16 years) performance score ≥ 40 at the time of study enrollment
4. Adequate organ function at the time of study enrollment as follows:

   * Bone marrow: ANC ≥ 1,000/μL, platelet count ≥ 100,000/μL (transfusion independent), hemoglobin concentration ≥ 8g/dL (may be transfused)
   * Renal: Serum creatinine concentration < 2x the institutional normal values for age or GFR > 70ml/min/1.73m2
   * Hepatic: Total bilirubin concentration < 1.5x the institutional upper limit of normal for age; SGPT < 5x the institutional upper limit of normal; albumin ≥ 2 g/dL
5. Electrocardiogram (EKG) with an average QTc interval < 450 msec. If a research participant has QTc interval ≥ 450 msec on screening EKG, the screening EKG may be repeated twice (at least 24 hours apart). The average QTc interval from the three screening EKGs must be < 450 msec in order for the research participant to be eligible for the study. Research participants with abnormal serum electrolytes and a QTc interval ≥ 450 msec should have a repeat EKG repeated once the concentration of serum electrolyte is corrected
6. Female research participants of childbearing age must not be pregnant (confirmed by serum or urine pregnancy test within 1 week of treatment start) or breast-feeding.
7. Female research participants of childbearing age and male research participants of child fathering potential must agree to use safe contraceptive methods

Exclusion Criteria:

1. Metastatic disease
2. Use of enzyme-inducing anticonvulsants
3. Research participants who received any other type of anticancer treatment
4. Research participants with uncontrolled infection
5. Research participants with any concomitant significant medical illness that in the investigator's opinion cannot be adequately controlled with appropriate therapy, or that would impair the evaluation of side effects related to this treatment, alter drug metabolism or the tolerance to this treatment
6. QTc interval prolongation with other medications that required discontinuation of that medication
7. Research participants with any history of cardiac arrhythmias or congenital long QT syndrome
8. Use of any concomitant medication that may cause QT interval prolongation and/or induce Torsades de Pointes
9. Hypertension defined as systolic and/or diastolic blood pressure > 95th percentile for age, height and gender, or blood pressure > 140/90 for research participants ≥ 18 years of age. If hypertension is detected, blood pressure values < 95th in two separate occasions need to be documented before registration. Body surface ≥ 1.8m2 for research participants enrolled on dosage levels 2, 3, and 4

Ages: 18 Months to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 25 (Actual)
Dates: Start 2009-10; Primary Completion 2012-04 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
To estimate the maximum tolerated dose (MTD) of the combination of vandetanib and dasatinib administered concurrently with RT in pediatric research participants with newly diagnosed DIPG | April 2012

SECONDARY OUTCOMES:
To determine the toxicities associated with the chronic use of vandetanib and dasatinib | July 2012
To characterize the pharmacokinetics of vandetanib and dasatinib in pediatric research participants | July 2012
To evaluate the influence of specific polymorphisms (e.g., CYP3A4/5) on the pharmacokinetics of vandetanib and dasatinib administered in combination | July 2012
To explore the association between plasma angiogenic factors and response to current therapy | July 2012
To evaluate the pharmacodynamics of dasatinib in target receptors and pathways in peripheral mononuclear cells | July 2012
To describe the research participants' and parents' perspective of the quality of life of children with newly diagnosed DIPG enrolled on this phase I trial | July 2012
To describe the quality of life of parents of pediatric research participants with newly diagnosed DIPG enrolled on this phase I trial | July 2012

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Broniscer, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols